CLINICAL TRIAL: NCT02329054
Title: Efficacy of Favipiravir in Reducing Mortality in Individuals With Ebola Virus Disease in Guinea
Brief Title: Efficacy of Favipiravir Against Ebola (JIKI)
Acronym: JIKI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C14-63
Record Dates: First submitted 2014-12-16; First posted 2014-12-31 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2015-03

CONDITIONS: Ebola Virus Disease
Keywords: Ebola Virus Disease; Antivirals; Mortality; Viral load; Proof-of-concept; Phase II trial; Guinea; Adults; Children
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — favipiravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Favipiravir (Experimental): Favipiravir (oral administration, 200 mg light yellow, round-shaped, coated divisible tablets that can be crushed and mixed with liquid)
  Interventions: Drug: Favipiravir

INTERVENTIONS:
Drug: Favipiravir — Group A1: Day-0 (inclusion), h0: 2400 mg; h8: 2400 mg; h16: 1200 mg. Day-1 to Day-9: 1200 mg bid.
  Group A2: Day-0 (inclusion), h0: 2400 mg; h8: 2400 mg; h16: 1200 mg. Day-1 to Day-9: 1200 mg bid.
  Group C: daily dosages will be adapted to their body weight.
  Other Names: AVIGAN

SUMMARY:
There is no specific treatment for Ebola Virus Disease (EVD). Current EVD care are supportive, and includes intravenous or oral rehydration, nutrition, pain killers, treatment of coinfections with antibacterial and antimalarial drugs, and blood transfusion when appropriate. Despite these interventions, mortality remains high since the ongoing Ebola outbreak in West Africa was declared in April.

Potential anti-Ebola specific interventions include convalescent plasma, monoclonal and polyclonal antibodies, small inhibitory RNA (siRNA), synthetic adenosine analogues or RNA polymerase inhibitors. All these interventions are considered investigational due to lack of data in humans with EVD.

In this study, the investigators chose to study the efficacy of favipiravir because this drug:

* showed anti-Ebola efficacy in immunodeficient murine models;
* has been studied in thousands of adult humans participating in anti-influenza trials, with good tolerance; it has been approved for treating novel or resistant influenza infections in Japan;
* is immediately available;
* can be used orally, and can be easily given in both adults and children because pills can be crushed and mixed in food or liquids;
* has recently been used in Europe for treating several patients with EVD; the French drug safety agency (ANSM) has reviewed published data as well as data provided by the firm (Toyama Chemical Co., Ltd), and approved its compassionate use in EVD.

Here the investigators propose to assess the efficacy of high-dosed favipiravir in reducing mortality in humans with EVD.

In the present trial "JIKI" (means "Hope" in "Kissi" language), investigators, sponsor, scientific advisory board and safety monitoring board will be coordinated in a very reactive way, so that any new fact can be discussed rapidly and the research plan can be adapted accordingly (change in drug dosage; use of drug combination; combination with another strategy such as passive immunization with convalescent plasma, etc.).

DETAILED DESCRIPTION:
Hypotheses:

1. The efficacy of antivirals in patients with EVD should correlate negatively with time since first symptoms. Thus, in this proof of concept trial, the main analysis will be done in adult patients with early symptoms in whom the efficacy is expected to be the highest;
2. Favipiravir for EVD should be given at higher doses than that previously tested in studies in human with influenza. For this trial, the dose was calculated based on pharmacokinetics simulations, to rapidly reach plasma concentrations associated with anti-EBOV activity.
3. A third assumption was made, given recent pre-trial data showing first a strong link between baseline viral load and mortality and second a higher mortality in children below 6 years: the efficacy of antivirals in patients with EVD should correlate negatively with viral load at start of treatment and with young age. Thus a secondary objective is the efficacy of favipiravir in adult patients and children >6 years with moderate baseline viral load (i.e. cycle threshold [Ct] ≥20 measured by RT-PCR) in whom the efficacy is expected to be the highest.

A comparative trial of favipiravir against a standard package of care (with or without placebo) has been deemed not appropriate because of: i) the highly sensitive social and political context; ii) the need to collect rapidly basic phase II evidence on the efficacy of high dosed favipiravir on EVD before choosing the best intervention(s) to be tested in phase III (favipiravir alone or in combination with other drugs; other therapeutic options including convalescent plasma).

Therefore, the investigators propose a non-comparative, proof-of-concept, phase II trial in patients with EVD, which will allow concluding within a few weeks:

* that mortality in patients starting favipiravir within 72 hours after the onset of first symptoms is inferior to mortality without treatment prior to the trial initiation;
* or that there is no trend that favipiravir brings significant benefit in terms of survival.

Objectives Primary objective: to assess the efficacy of high-dosed favipiravir in reducing mortality in humans with EVD.

Secondary objectives: to assess the evolution of EBOV plasma RNA and infectious loads under treatment; the tolerance of favipiravir; the viral micro-diversity of EBOV, the trough concentrations of favipiravir and factors associated with mortality and toxicity.

Groups In this protocol, the investigators will refer to the following groups according to age and duration of symptoms*: Group A1: adults with time between first symptoms and first dose of favipiravir ≤72h; Group A2: adults with time between first symptoms and first dose of favipiravir >72h and Group C: all children >1 year and weighting ≥10kg. Time of first symptom refers to the time of the beginning of any symptom considered to be related to EVD.

* Symptoms to be considered will be: acute onset of fever, severe headache, myalgia, extreme fatigue, vomiting, diarrhoea, abdominal pain, or unexplained hemorrhage.

Given recent pre-trial data, a second definition of groups was also used: group AC1: adults and children >6 years with baseline Ct ≥20; group AC2: adults and children >6 years with baseline Ct values <20; group YC: young children ≤6 years and >1 year.

Sample size: recruitment in the trial will be kept opened in all groups until group A1 reaches 60 participants, unless early termination is recommended by the DSMB. Because we expect the efficacy of the treatment to be the maximum in patients with early symptoms, the sample size calculation was based on the analysis of mortality in group A1.

The observed pre-trial mortality was estimated using the three months data (from 15/08/2014 to 15/11/2014) of the MSF database in the Gueckedou EVD centre. Given those estimations, and to remain pragmatic and conservative, we set the pre-trial mortality to 55% for groups A1, A2, C.

With 60 participants in group A1, the power to conclude that mortality in the trial will be -20% inferior to pre-trial mortality will be equal to 89%.

Statistical analysis for primary outcome: mortality by Day-14 with 95% CI will be reported overall and in each group separately. Day-0 is the day of the first dose of favipiravir.

In group A1, if the number of deaths is <24 (40%) out of 60 participants, the upper bound of the 95%CI will be <55%.

In group A2, if the number of deaths is <54 (45%) out of 120 participants, the upper bound of the 95%CI will be <55%.

In group C, if the number of deaths is <17 (38%) out of 45 participants, the upper bound of the 95%CI will be <55% In each group (A1, A2, C), the investigator will conclude that favipiravir decreases mortality if the upper bound of the 95% CI does not include the observed pre-trial mortality (55%) in untreated patients with same duration of symptoms prior to trial initiation.

Statistical analysis for secondary outcomes: mortality by Day-14 with exact 95%CI will be reported according to the second group definition (AC1, AC2, YC). In each group, we will conclude that favipiravir decreases mortality if the upper bound of the 95% CI does not include the observed pre-trial mortality (30%, 85% and 70%, respectively) in untreated patients with same characteristics prior to trial initiation.

All the following outcomes will be analysed overall and separately by the two group definitions (A1, A2, C or AC1, AC2, YC): the evolution of EBOV plasma RNA and infectious loads between Day-0 and the end of follow up will be described in each patient. The numbers, proportions and exact 95% CI will be described for grade 3-4 adverse events; resistance mutations; and patients reaching criteria for cure at Day-30. The distribution (median, IQR, min-max) of initial and maximal viral load, time to maximal viral load and to undetectability, and rate of increase/decrease will be reported. The distribution of trough concentrations of favipiravir at each point and the inter- and intra-patient variability of concentrations will be described.

Factors associated with mortality by Day-14, cure at Day-30 and grade 3-4 clinical or biological adverse events (including time between first symptoms and treatment initiation, evolution of EBOV viral load, trough concentrations of favipiravir) will be studied.

Stopping rules for futility: there will be intermediate analyses of mortality for futility only, performed every 20 adults in each group and every 10 children:

* Adults: recruitment in the two groups A1 and A2 will be prematurely stopped if the results show that the trial is unlikely to prove that mortality with favipiravir is <55%;
* Children: recruitment in the group C will be prematurely stopped if the results show that the trial is unlikely to prove that mortality with favipiravir is <55%.

Toxicity: deaths will be reported to the sponsor and to the DSMB on a daily basis; SAE other than death will be reported to the sponsor and to the DSMB on a weekly basis.

Sponsor and coordination The trial sponsor is the INSERM. The international coordinating, monitoring and data management centre will be the "Mereva" clinical trial unit (CTU), an international team with members affiliated to the Inserm 897 Unit, University of Bordeaux and to the "Pacci/ANRS" research site in Abidjan. Trial coordinating, monitoring and data management activities will be coordinated by an International Clinical Project Manager (CPM). In Guinea, where the trial will be conducted, a trial country coordination center (CCC) will be put in place, lead by a country CPM who will work in close collaboration with the international CPM and with the participating clinical centres.

The trial will be conducted and monitored according to a Standard Operating Procedures (SOPs) manual.

Monitoring

In order to ensure the clinical trial is conducted properly, the CTU and CCC will coordinate all study activities of the Project Team. This includes in particular to:

* Set up and monitor workflows, timelines, milestones and tracking tools;
* Conduct regular team meetings to discuss project status, activities, and address issues;
* Maintain daily contact with principal investigators, sponsor and clinical sites;
* Provide status reports to principal investigator, DSMB, and SAB;
* Support the study sites with study related questions;
* Ensure that study drug is being stored, dispensed, and accounted for according to specifications;
* Check the completeness of patient records, the accuracy of entries in the database, the adherence to the protocol, SOPs and to Good Clinical Practice. Monitoring standards require full verification for the presence of informed consent, adherence to the inclusion/exclusion criteria, documentation of serious adverse events (SAEs), and the recording of data that will be used for all primary and safety variables.

The investigator must give the CCC access to all relevant source documents to confirm their consistency with the CRF and database entries. For this particular trial, some documents filed in within the isolation ward will have to be destroyed in order to avoid contamination. Data recorded on a document that will have to be destroyed will be defined before study start.

the investigators put particular focus on structured communication, and, together with the principal investigators and the partners, will define the communication plan which includes the key communication areas such as meetings, trainings, telephone conferences, internal project meetings, monitoring plan meetings and report updates.

Investigators at each clinical site will keep a hard copy of the Trial Master File (TMF), containing all essential technical (protocol, SOPs, etc.), and regulatory (insurance, IRB approvals, task delegation descriptions, bio-sketches, agreements, etc.) trial documents. The country CPM will be responsible for checking that the files containing the hard copy of the TMF documents at each trial clinic and at the CCC are up-to-date. All TMF documents will also be made available online to investigators on a private website ("eTMF"). The international CPM will be responsible for routinely updating the documentation on the trial website.

Data management

The CTU will develop by December 1st, 2014:

A case report form (CRF): data will be collected on hard copy CRF. The medical investigator or his/her designated representative will be responsible for filling out the forms.

A database: Data will be entered online in a system that will ensure data encryption, restricted access to the database, daily back-up, and tracking of edits.

A Data Management Plan (DMP) and Data Validation Plan (DVP), including the quality control process to ensure completeness, validity, consistency, timeliness and accuracy.

Training will be provided to all members of the study team involved in data collection data entry, data check and monitoring.

The CTU data managing team will conduct data review and handle queries on a weekly basis, and reconcile the safety database with the clinical database.

ELIGIBILITY:
Inclusion Criteria:

* age >1 year and weighting ≥10kg,
* EVD confirmed by a positive qualitative PCR test,
* signed informed consent (signed by the parents/adults guardians in case of minor patient).

Non inclusion-criteria:

* pregnancy*,
* inability to take the drug (encephalopathy, severe vomiting). * Emergency use of favipiravir in pregnant women outside of the trial is envisaged and under evaluation.

In this protocol, the investigators will refer to the following groups according to age and duration of symptoms**:

* Group A1: adults with time between first symptoms and first dose of favipiravir ≤72h;
* Group A2: adults with time between first symptoms and first dose of favipiravir >72h;
* Group C: all children >1 year and weighting ≥10kg. Time of first symptom refers to the time of the beginning of any symptom considered to be related to EVD. **Symptoms to be considered will be: acute onset of fever, severe headache, myalgia, extreme fatigue, vomiting, diarrhoea, abdominal pain, or unexplained hemorrhage.

The division in groups is a matter of analysis, and will not be perceptible by the patients during the trial process. Patients in the three groups will receive the same treatment and will be followed under the same procedures, with only two exceptions: the number of additional blood sample collections will be lower in group A2 and C (n=2) than in group A1 (n=3) and daily dosages will be adapted to the body weight in group C.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Mortality | Day-14
  Day-0 is the day of the first dose of favipiravir

SECONDARY OUTCOMES:
Evolution of EBOV plasma RNA and infectious loads | routine care venepuncture (Day-0; end of symptoms (EOS)+72h and EOS+96h if EOS >Day-9; or Day-12 and Day-13 if EOS <Day-9); (ii) additional trial venepuncture at: Day-2, Day-4 and Day-30 in group A1; Day-2 and Day-30 in group A2
Occurrence of grade 3 or 4 clinical or biological adverse events (Common Terminology Criteria for Adverse Events, CTAE, v3.0) | participants will be followed for the duration of hospital stay up to Day-14
Evolution of viral micro-diversity of EBOV (including potential resistance mutations) | routine care venepuncture (Day-0; end of symptoms (EOS)+72h and EOS+96h if EOS >Day-9; or Day-12 and Day-13 if EOS <Day-9); (ii) additional trial venepuncture at: Day-2, Day-4 and Day-30 in group A1; Day-2 and Day-30 in group A2
Plasma trough concentrations of favipiravir | routine care venepuncture (Day-0; end of symptoms (EOS)+72h and EOS+96h if EOS >Day-9; or Day-12 and Day-13 if EOS <Day-9); (ii) additional trial venepuncture at: Day-2, Day-4 and Day-30 in group A1; Day-2 and Day-30 in group A2
Criteria for cure | Day-30
  Composite criteria for cure are the following:
  * 4 days without fever or significant symptoms AND;
  * able to feed and walk independently AND;
  * two consecutive negative qualitative PCR.
Mortality | Day-14 according to the second group definition (AC1, AC2, YC)
  Day-0 is the day of the first dose of favipiravir

CONTACTS AND LOCATIONS:
Overall Officials: Denis Malvy, Professor, Principal Investigator — CHU de Bordeaux & INSERM, Université de Bordeaux, France
Locations (4):
- Guinea (4):
  - The caregivers treatment center, Conakry
  - MSF Ebola treatment centre, Gueckedou
  - French Red Cross Ebola care center, Macenta
  - ALIMA Ebola care center, Nzérékoré

REFERENCES:
- [Background] Mentre F, Taburet AM, Guedj J, Anglaret X, Keita S, de Lamballerie X, Malvy D. Dose regimen of favipiravir for Ebola virus disease. Lancet Infect Dis. 2015 Feb;15(2):150-1. doi: 10.1016/S1473-3099(14)71047-3. Epub 2014 Nov 28. No abstract available. PMID 25435054
- [Result] Nguyen TH, Guedj J, Anglaret X, Laouenan C, Madelain V, Taburet AM, Baize S, Sissoko D, Pastorino B, Rodallec A, Piorkowski G, Carazo S, Conde MN, Gala JL, Bore JA, Carbonnelle C, Jacquot F, Raoul H, Malvy D, de Lamballerie X, Mentre F; JIKI study group. Favipiravir pharmacokinetics in Ebola-Infected patients of the JIKI trial reveals concentrations lower than targeted. PLoS Negl Trop Dis. 2017 Feb 23;11(2):e0005389. doi: 10.1371/journal.pntd.0005389. eCollection 2017 Feb. PMID 28231247
- [Result] Eloy P, Laouenan C, Beavogui AH, Keita S, Manchon P, Etard JF, Sissoko D, Mentre F, Malvy D. High doses of favipiravir in two men survivors of Ebola virus disease carrying Ebola virus in semen in Guinea. IDCases. 2022 Jan 21;27:e01412. doi: 10.1016/j.idcr.2022.e01412. eCollection 2022. PMID 35127447
- [Result] Sissoko D, Laouenan C, Folkesson E, M'Lebing AB, Beavogui AH, Baize S, Camara AM, Maes P, Shepherd S, Danel C, Carazo S, Conde MN, Gala JL, Colin G, Savini H, Bore JA, Le Marcis F, Koundouno FR, Petitjean F, Lamah MC, Diederich S, Tounkara A, Poelart G, Berbain E, Dindart JM, Duraffour S, Lefevre A, Leno T, Peyrouset O, Irenge L, Bangoura N, Palich R, Hinzmann J, Kraus A, Barry TS, Berette S, Bongono A, Camara MS, Munoz VC, Doumbouya L, Harouna S, Kighoma PM, Koundouno FR, Lolamou R, Loua CM, Massala V, Moumouni K, Provost C, Samake N, Sekou C, Soumah A, Arnould I, Komano MS, Gustin L, Berutto C, Camara D, Camara FS, Colpaert J, Delamou L, Jansson L, Kourouma E, Loua M, Malme K, Manfrin E, Maomou A, Milinouno A, Ombelet S, Sidiboun AY, Verreckt I, Yombouno P, Bocquin A, Carbonnelle C, Carmoi T, Frange P, Mely S, Nguyen VK, Pannetier D, Taburet AM, Treluyer JM, Kolie J, Moh R, Gonzalez MC, Kuisma E, Liedigk B, Ngabo D, Rudolf M, Thom R, Kerber R, Gabriel M, Di Caro A, Wolfel R, Badir J, Bentahir M, Deccache Y, Dumont C, Durant JF, El Bakkouri K, Uwamahoro MG, Smits B, Toufik N, Van Cauwenberghe S, Ezzedine K, D'Ortenzio E, Pizarro L, Etienne A, Guedj J, Fizet A, de Sainte Fare EB, Murgue B, Tran-Minh T, Rapp C, Piguet P, Poncin M, Draguez B, Duverger TA, Barbe S, Baret G, Defourny I, Carroll M, Raoul H, Augier A, Eholie SP, Yazdanpanah Y, Levy-Marchal C, Antierrens A, Van Herp M, Gunther S, de Lamballerie X, Keita S, Mentre F, Anglaret X, Malvy D; JIKI Study Group. Correction: Experimental Treatment with Favipiravir for Ebola Virus Disease (the JIKI Trial): A Historically Controlled, Single-Arm Proof-of-Concept Trial in Guinea. PLoS Med. 2016 Apr 5;13(4):e1002009. doi: 10.1371/journal.pmed.1002009. eCollection 2016 Apr. PMID 27046271
- [Derived] Sissoko D, Laouenan C, Folkesson E, M'Lebing AB, Beavogui AH, Baize S, Camara AM, Maes P, Shepherd S, Danel C, Carazo S, Conde MN, Gala JL, Colin G, Savini H, Bore JA, Le Marcis F, Koundouno FR, Petitjean F, Lamah MC, Diederich S, Tounkara A, Poelart G, Berbain E, Dindart JM, Duraffour S, Lefevre A, Leno T, Peyrouset O, Irenge L, Bangoura N, Palich R, Hinzmann J, Kraus A, Barry TS, Berette S, Bongono A, Camara MS, Chanfreau Munoz V, Doumbouya L, Souley Harouna, Kighoma PM, Koundouno FR, Rene Lolamou, Loua CM, Massala V, Moumouni K, Provost C, Samake N, Sekou C, Soumah A, Arnould I, Komano MS, Gustin L, Berutto C, Camara D, Camara FS, Colpaert J, Delamou L, Jansson L, Kourouma E, Loua M, Malme K, Manfrin E, Maomou A, Milinouno A, Ombelet S, Sidiboun AY, Verreckt I, Yombouno P, Bocquin A, Carbonnelle C, Carmoi T, Frange P, Mely S, Nguyen VK, Pannetier D, Taburet AM, Treluyer JM, Kolie J, Moh R, Gonzalez MC, Kuisma E, Liedigk B, Ngabo D, Rudolf M, Thom R, Kerber R, Gabriel M, Di Caro A, Wolfel R, Badir J, Bentahir M, Deccache Y, Dumont C, Durant JF, El Bakkouri K, Gasasira Uwamahoro M, Smits B, Toufik N, Van Cauwenberghe S, Ezzedine K, D'Ortenzio E, Pizarro L, Etienne A, Guedj J, Fizet A, Barte de Sainte Fare E, Murgue B, Tran-Minh T, Rapp C, Piguet P, Poncin M, Draguez B, Allaford Duverger T, Barbe S, Baret G, Defourny I, Carroll M, Raoul H, Augier A, Eholie SP, Yazdanpanah Y, Levy-Marchal C, Antierrens A, Van Herp M, Gunther S, de Lamballerie X, Keita S, Mentre F, Anglaret X, Malvy D; JIKI Study Group. Experimental Treatment with Favipiravir for Ebola Virus Disease (the JIKI Trial): A Historically Controlled, Single-Arm Proof-of-Concept Trial in Guinea. PLoS Med. 2016 Mar 1;13(3):e1001967. doi: 10.1371/journal.pmed.1001967. eCollection 2016 Mar. PMID 26930627